CLINICAL TRIAL: NCT04549831
Title: Identification of the Genetic Bases Determining COVID-19 Clinical Variability in the Italian Population
Brief Title: Genetic Bases of COVID-19 Clinical Variability
Acronym: GEN-COVID
Status: Recruiting | Type: Observational
Sponsor: University of Siena (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Ospedale San Donato, Arezzo (Unknown); Ospedale della Misericordia (Other); Azienda Ospedaliera Ospedale Maggiore di Crema (Other); University of Modena and Reggio Emilia (Other); ASST Fatebenefratelli Sacco (Other); Azienda Ospedaliera di Perugia (Other); Ospedale dell'Angelo, Venezia-Mestre (Other); Azienda Ulss 2 Marca Trevigiana (Other); Cardarelli Hospital (Other); Azienda Ospedaliera dei Colli (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); Istituto Giannina Gaslini (Other); Istituti Ospitalieri di Cremona (Other); IRCSS Lazzaro Spallanzani, Roma (Unknown); ASST Santi Paolo e Carlo (Other); ASST Valtellina e Alto Lario (Unknown); Azienda USL Toscana Sud Est (Other Government); ULSS1 Dolomiti, Belluno (Unknown); Asst Degli Spedali Civili Di Brescia (Other); IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo (Unknown); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Ospedale Luigi Curto, Polla (Unknown); Istituto Auxologico Italiano (Other); CEINGE Biotecnologie Avanzate, Napoli (Unknown)
Responsible Party: Principal Investigator, Francesca Mari, Principal Investigator, Azienda Ospedaliera Universitaria Senese
Other Study IDs: 16917
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Host Genetics; Genetic susceptibility
MeSH Terms: conditions — COVID-19; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and derivates such as plasma, serum, DNA, lymphocytes, lymphoblastic cell lines, naso/oro-pharyngeal swab and derivates such as RNA, DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 PCR positive individuals: Adult (> o equal to 18 years) SARS-CoV-2 PCR positive individuals with different clinical outcome: from asymptomatic to severely affected COVID-19 patients.
  Interventions: Genetic: Massive parallel sequencing of host genome

INTERVENTIONS:
Genetic: Massive parallel sequencing of host genome — Massive parallel sequencing and genotyping of host genome of individuals infected with SARS-CoV-2 and showing different clinical outcomes from asymptomatic to severely affected patients in order to identify the genetic determinants of severe COVID-19 and the genetic protective factors.

SUMMARY:
GEN-COVID multicenter study aims to identify the genetic variants of the host genome responsible for the clinical variability of patients with COVID-19. This variability to date is only partially related to the age and comorbidities of patients. The primary objective of the study is therefore to identify genetic variants associated with the severity of the disease, while the secondary objective consists in the identification of variants associated with longitudinal disease trajectories.

This is a laboratory study that involves the conduct of genetic investigations, including whole exome sequencing and genome wide association studies, on human biological material from patients affected by COVID-19.

Clinical information useful to describe the level of disease severity will be also collected for each enrolled patient.

A total of at least 2,000 COVID-19 patients is expected to be included.

DETAILED DESCRIPTION:
The outbreak of the coronavirus disease 2019 (COVID-19), the Severe Acute Respiratory Syndrome caused by SARS-CoV-2, that first appeared in December 2019 in Wuhan, Huanan, Hubei Province of China, has resulted in millions of cases worldwide within a few short months, and rapidly evolving into a real pandemic. The COVID-19 pandemic represents an enormous challenge to the world's healthcare systems. Among the European countries, Italy was the first to experience the epidemic wave of SARS-CoV-2 infection, accompanied by a severe clinical picture and a mortality rate reaching 14%.

The disease is characterized by a highly heterogeneous phenotypic response to SARS-CoV-2 infection, with the large majority of infected individuals having only mild or even no symptoms. However, the severe cases can rapidly evolve towards a critical respiratory distress syndrome and multiple organ failure. The symptoms of COVID-19 range from fever, cough, sore throat, congestion, and fatigue to shortness of breath, hemoptysis, pneumonia followed by respiratory disorders and septic shocks.

The GEN-COVID is a multicentre academic observational study designed to collect and systematize biological samples and clinical data across multiple hospitals and healthcare facilities in Italy with the purpose of deriving patient-level phenotypic and genotypic data. The project aims to identify the genetic determinants of COVID-19 clinical variability studying host genetics. Genetic analyses will include Genome Wide Association Studies, performed by the Institute of Molecular Medicine in Finland (FIMM), and Whole Exome Sequencing (WES) performed by the University of Siena. SARS-CoV-2 infected individuals (swab virus PCR-positive) showing clinical different severity will be collected. In particular enrolled subjects will include only adults (subjects with age higher or equal to 18 years) with the following clinical status types: asymptomatic individuals, home care patients with mild symptoms and hospitalized patients (i-those requiring invasive ventilation; ii-those requiring non-invasive ventilation i.e. CPAP and BiPAP, and high-flows oxygen therapy; iii- those requiring conventional oxygen therapy, and iv-those not requiring oxygen therapy).

Funding. MIUR project "Dipartimenti di Eccellenza 2018-2020" to Department of Medical Biotechnologies University of Siena, Italy; Private donors for COVID research (Italian D.L. n.18 March 17, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18
* SARS-CoV-2 PCR positive on swab

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients, outpatients, asymptomatic individuals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
To identify the genetic determinants of COVID-19 severity | 6 years
  Identification of one or more candidate gene(s) responsible for the severe outcome and subsequent use of it/them for prognostic purposes and preventive treatment and/or care.

SECONDARY OUTCOMES:
To identify the genetic determinants of COVID-19 clinical trajectories. | 6 years
  Identification of candidate gene(s) responsible for the COVID-19 clinical trajectories.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Mari, MD, PhD, Principal Investigator — University of Siena
Locations (1):
- University of Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: Yes
Relevant information coming from the genetic results of the study will be made available to the scientific community through the Network of Italian Genomes (NIG)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Already available
Access Criteria: Publicly available
URL: http://nigdb.cineca.it

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Derived] Bergantini L, Baldassarri M, d'Alessandro M, Brunelli G, Fabbri G, Zguro K, Degl'Innocenti A; GEN-COVID Multicenter study; Fallerini C, Bargagli E, Renieri A. Ultra-rare RTEL1 gene variants associate with acute severity of COVID-19 and evolution to pulmonary fibrosis as a specific long COVID disorder. Respir Res. 2023 Jun 16;24(1):158. doi: 10.1186/s12931-023-02458-7. PMID 37328761
- [Derived] Fallerini C, Daga S, Mantovani S, Benetti E, Picchiotti N, Francisci D, Paciosi F, Schiaroli E, Baldassarri M, Fava F, Palmieri M, Ludovisi S, Castelli F, Quiros-Roldan E, Vaghi M, Rusconi S, Siano M, Bandini M, Spiga O, Capitani K, Furini S, Mari F; GEN-COVID Multicenter Study; Renieri A, Mondelli MU, Frullanti E. Association of Toll-like receptor 7 variants with life-threatening COVID-19 disease in males: findings from a nested case-control study. Elife. 2021 Mar 2;10:e67569. doi: 10.7554/eLife.67569. PMID 33650967
- See also: Employing a Systematic Approach to Biobanking and Analyzing Genetic and Clinical Data for Advancing COVID-19 Research — http://doi.org/10.1101/2020.07.24.20161307
- See also: GEN-COVID: Impact of Host Genome on COVID-19 clinical variability — http://sites.google.com/dbm.unisi.it/gen-covid